CLINICAL TRIAL: NCT04239963
Title: Behavioral and Electrophysiological Effects of Ketamine in Treatment-Resistant Depression
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Diego Pizzagalli, Director, Center for Depression, Anxiety and Stress Research, Mclean Hospital
Other Study IDs: 2019P003371
Record Dates: First submitted 2020-01-15; First posted 2020-01-27 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Controls: Subjects who have no history of clinical depression or other psychological disorder
- Current MDD: Subjects experiencing a current episode of Major Depressive Disorder.

SUMMARY:
The overarching goal of the present study is to evaluate the effect of a subanesthetic dose of ketamine 24-hour post-injection on resting state functional connectivity, cognitive control, and reward learning.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) participants with treatment-resistant depression (TRD) will be recruited from McLean's Ketamine clinic. Suitability for Ketamine treatment will be determined as typically done by the service - through evaluation by the clinicians on the staff of the Ketamine Service who perform psychiatric consultations and assessments for Ketamine suitability. Potential subjects will be informed about the study only after they have received a positive consultation at the clinic and have already agreed to receive the treatment.

This study consists of a set of questionnaires, urine drug screen, and electroencephalogram (EEG) recordings.

ELIGIBILITY:
Inclusion Criteria (MDD Subjects):

* All genders, races, and ethnic origins, aged between 18 and 70;
* DSM-5 diagnostic criteria for MDD (diagnosed with the use of the Structured Clinical Interview for DSM-5 (SCID-5));
* A score of ≥32 on the Inventory of Depressive Symptomatology-Clinician Rated (IDS-C30).
* Capable of providing written informed consent, and fluent in English;
* Right-handed;
* Treatment Resistant (as assessed using the MGH Antidepressant Response Questionnaire)
* Have already decided to receive ketamine treatment as part of their standard clinical care

Inclusion Criteria (Control Subjects):

* All genders, races, and ethnic origins, aged between 18 and 70;
* Absence of medical, neurological, and psychiatric illness (including alcohol and substance abuse), as assessed by subject history and a structured clinical interview (SCID-I/NP);
* A baseline Quick Inventory of Depressive Symptomatology (QIDS) score ≤ 5;
* A baseline Hamilton Depression Rating Scale (HDRS) score ≤ 7;
* Capable of providing written informed consent, and fluent in English;
* Right-handed;
* No first-degree relative with mood or psychotic disorder.

Exclusion Criteria (All Subjects):

* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease;
* History of seizure disorder;
* History or current diagnosis of any of the following DSM-5 psychiatric illnesses: schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, substance abuse disorder;
* Clinical or laboratory evidence of hypothyroidism, hyperthyroidism, or other thyroid disorder that is not controlled by medication;
* Substance use assessed by physician as dangerous for ketamine treatment;
* Untreated glaucoma;
* Complex post-traumatic stress disorder (PTSD) with dissociation;
* Patients with a lifetime history of electroconvulsive therapy (ECT).
* Participants with a lifetime history of ketamine use.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to recruit 30 TRD individuals with current MDD without psychotic features and 30 demographically matched healthy controls. All participants will be ketamine-naïve.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Feedback-related positivity (FRP) amplitudes over frontocentral scalp regions in response to rewarded trials versus no-reward trials | Baseline
  Relative FRP response is the primary outcome measure for the probabilistic reward task (PRT).
Event-related negativity (ERN) amplitudes over frontocentral scalp regions in response to correct trials versus incorrect trials. | Baseline
  Relative ERN response is the primary outcome measure for the flanker task.
Behavioral Performance on the Probabilistic Reward Task (PRT) | Baseline
  The Probablilistic Reward Task operationalizes positive reinforcement learning
Behavioral Performance on the Flanker Task | Baseline
  The Flanker Task is a cognitive task that measures response inhibition to assess the ability to suppress responses that are inappropriate in a particular context.
Rumination | Baseline
  Severity of rumination will be assessed using the Rumination Response Scale (RRS). The RRS has a minimum score of 22 and a maximum score of 88. Higher scores indicate higher degrees of ruminative symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Pizzagalli, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States